CLINICAL TRIAL: NCT06795867
Title: Does Acceptance and Commitment Therapy (ACT) Improve Disability in Chronic Migraine? A Randomized Headache Center Trial
Brief Title: Acceptance and Commitment Therapy to Improve Disability in Chronic Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Paul B. Rizzoli, M.D., Division Chief, Headache, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P002621
Record Dates: First submitted 2025-01-14; First posted 2025-01-28 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Chronic Migraine
Keywords: migraine; chronic migraine; behavioral management; acceptance and commitment therapy
MeSH Terms: conditions — Migraine Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT plus usual treatment (Active Comparator): the addition of acceptance and commitment therapy to usual treatment
  Interventions: Behavioral: acceptance and commitment therapy
- Usual treatment alone (No Intervention): usual treatment without additional intervention

INTERVENTIONS:
Behavioral: acceptance and commitment therapy — a 'third wave behavioral management
  Arms: ACT plus usual treatment

SUMMARY:
The goal of this clinical trial is to learn if the behavioral treatment called Acceptance and Commitment Therapy (ACT) works to improve disability in adults with chronic migraine. The main questions it aims to answer are:

Does the use of ACT added to usual treatment improve scores on questionnaires designed to measure daily functioning and activity? Does the use of ACT added to usual treatment improve scores on diaries designed to measure headache frequency and pain?

Researchers will compare adding ACT to usual headache treatments to usual headache treatments without ACT.

Participants who are selected for ACT will take 8 classes to learn ACT and then will practice it at home, in addition to their regular headache treatment. Those not selected will continue their regular headache treatment. Four times over the following year, participants will answer questions about their symptoms during each of four virtual visits. They will also keep a daily headache diary during the study

DETAILED DESCRIPTION:
Background and Significance

Chronic migraine prevalence is 3% of the migraine population, though the majority of patients seen in a headache center and is often a disabling condition. Pharmacologic management has expanded and improved in recent years though it nonetheless provides incomplete control in many patients. Even the best specialty headache clinic management falls short in providing relief to some chronic migraine patients. Behavioral therapies have shown efficacy in pain conditions, including migraine. Behavioral treatments may improve disability related to headache more so than headache days, a traditional measure of headache treatment efficacy. However, reduced disability is, in the end, the most important outcome in headache management. If behavioral management, in addition to usual treatment, can improve disability outcomes in patients, an argument can be made for expanding access to these modalities in the headache clinic setting.

Acceptance & Commitment Therapy (ACT), often referred to as the "third wave of cognitive behavioral approaches," has helped treat a variety of conditions, including depression, anxiety, and chronic non-headache pain. ACT departs from mainstream cognitive behavioral therapy approaches in a number of respects. The most unique aspect is learning to accept one's present condition (vs. the more typical approaches that focus on direct approaches for managing and coping with a given condition). The overarching aim of ACT-based therapies for pain is to promote greater psychological flexibility by cultivating six different positive psychological capacities: acceptance, defusion, mindfulness, sense of self, values, and committed actions. Acceptance in ACT is not merely tolerance: rather, it is the active and nonjudgmental embracing of experiences in the here and now as they are. Mindfulness is one of the ways to increase acceptance, achieve cognitive defusion and thus increase behavioral flexibility. Studies have documented the effectiveness of ACT interventions for improving disability, lessening the impact of pain, and developing resilience for varied types of recurrent non-headache pain conditions and migraine. The latter finding is particularly important as individuals with low resilience, especially those currently experiencing chronic pain, are more susceptible to emotional difficulties when exposed to stressful situations and this, in turn, gives rise to conditions such as depression or anxiety.

Studies examining the clinical utility of mindfulness and ACT in chronic pain conditions and migraine have demonstrated how these practices help by increasing pain tolerance, reducing the need for symptomatic medications, reducing the frequency of migraine attacks as well as the course of migraine episodes, and by modulating certain personality characteristics of patients with migraine, such as anxiety, rigidity, low acceptance, and low resilience. Patients with pain can be effectively supported by nonpharmacological approaches, such as ACT, to manage their pain and the anxiety connected to pain, by improving their clinical condition, and by decreasing the likelihood of a long-term negative course. Specifically, patients with chronic migraine may benefit from attending ACT treatment not only in terms of clinical improvement, but also through reduction of the medication intake. The integration of ACT into standard care merits continued study, replication and extension to other sites to more fully identify both the strengths and limitations of this particular integrative approach

Hypothesis: The addition of Acceptance and Commitment Therapy to usual care will improve measures of disability in chronic migraine participants, as measured by the Headache Disability Index, comparing changes in scores from baseline to 3 months. Secondary and exploratory analyses are as noted. This is a single site randomized, open-label phase II pilot study. Participants will be randomized 1:1 with the following method using a computerized random generator into 2 groups: ACT and usual treatment. Initial ACT training requires 8 virtual group visits over 2 months. All participants will be assessed at 3, 6 and 12 months. ACT training involves 8 one-hour sessions covering six different positive psychological capacities: acceptance, defusion, mindfulness, sense of self, values, and committed actions, followed by two review sessions. The goal of ACT is to improve mindfulness. Mindfulness is one of the ways to increase acceptance, achieve cognitive defusion and thus increase behavioral flexibility which should lead to reduced disability in the migraine population.

Chronic migraine is a potentially disabling condition that requires medical management in most patients. Studying chronic migraine patients without the use of some form of standard or usual medical management would not be feasible. Restricting usual management would be unduly harsh and would limit recruitment. Thus, both groups will be offered usual or standard management. Conversely it seems clear that medical management is not a complete solution in many patients. Though many patients improve with usual treatment, many still report some level of disability. This study tests the hypothesis that ACT can improve reported disability in these patients.

A participant is considered to have completed the study if he or she has completed the baseline assessment, ACT training if so randomized and the 3-month, 6-month and 12-month follow-up assessments. Participants will be allowed to miss up to 2 sessions and miss 0 visits in order to continue in the study.

After the consent process is completed, the participant will be randomized to group A or B and questionnaires will be administered.

Three or four training groups of 5 participants each are anticipated. Intervention attendance will be monitored and recorded. Training is conducted by a physician experienced in the procedure and is based on a prior published protocol.

The intervention will be completed virtually, and no in-person offerings are anticipated. The intervention will be done by a study team psychologist trained in the use of ACT. Each session has a theme as noted in the included training documents. Intervention sessions will not be recorded. Subjects may interact during the training meetings.

This is an open-label trial. Patients will be randomized to receive either ACT or usual treatment. Randomization will use a permuted block method. The randomization ratio will be 1:1. A biostatistician will generate the randomization codes and upload the randomization list in the Redcap system.

In addition, participants will maintain daily diaries on paper and this data will be collected periodically. These will be used to measure abortive medication intake and practice times.

Regular, daily or near-daily, practice of mindfulness both during and after the intervention sessions will be encouraged. Practice may be recorded in the daily diaries that participants are encouraged to maintain.

The data to be collected at the time of study intervention discontinuation will include the following:

* The reason(s) for discontinuing the participant from the intervention, and methods for determining the need to discontinue
* If the participant is due to complete assessments within 2 weeks of being discontinued from the study intervention, those assessments will be administered at the time of discontinuation; if the next scheduled assessments are more than 2 weeks from the discontinuation date, the discontinued participant will wait for the next scheduled assessment. Thereafter, the participant will be included in all future scheduled assessments, even though not participating in the intervention.

Participants are free to withdraw from participation in the study at any time upon request.

An investigator may discontinue a participant from the study for the following reasons:

* Significant study intervention non-compliance
* Lost-to-follow up; unable to contact subject (see Section 7.3, Lost to Follow-Up)
* Any event or medical condition or situation occurs such that continued collection of follow-up study data would not be in the best interest of the participant or might require an additional treatment that would confound the interpretation of the study
* The participant meets an exclusion criterion (either newly developed or not previously recognized) that precludes further study participation

The reason for participant discontinuation or withdrawal from the study will be recorded on the Case Report Form (CRF). Subjects who sign the informed consent form and are randomized but do not receive the study intervention may be replaced. Subjects who sign the informed consent form, and are randomized and receive the study intervention, and subsequently withdraw, or are discontinued from the study will not be replaced.

A participant will be considered lost to follow-up if he or she fails to return for one scheduled visit and study staff are unable to contact the participant after at least 3 attempts.

Study procedures as per the Schedule of Activities, include questionnaires and the recording of diary information, along with assessment of any adverse events:

Data will be maintained in a secure fashion as described elsewhere in the protocol.

No specific provision is allowed for transmittal of specific questionnaire results to participants since individual scores are not likely to be of value to the participant.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to engage in the consent process
* Willingness to participate in the study, despite randomization outcome
* Availability for the duration of the study
* Diagnosis of chronic migraine followed at the Graham Headache Center
* Access to the necessary resources for participating in a technology-based intervention

Exclusion Criteria:

* Known major depression or other psychiatric condition
* Non-English speaking
* Secondary headache diagnosis
* Psychotherapy in the prior 18 months
* Any reason the provider feels would limit participant ability to learn or practice ACT
* Any previous experience with mindfulness or meditation approaches

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in Headache Disability Index | 3 months
  Change in Headache Disability Index from baseline to 3 months. Scores at 3 months minus scores at baseline.

SECONDARY OUTCOMES:
Disability Measures | Baseline, 3,6 and 12 months
  Headache Disability Index.
Anxiety Assessment | Baseline, 3, 6 and 12 months
  Hospital Anxiety and Depression Scale
Catastrophizing Score | Baseline, 3, 6 and 12 months
  Patient Catastrophizing Scale
Mindfulness Assessment | Baseline, 3, 6 and 12 months
  Five Facet Mindfulness Questionnaire
Disability Measures | Baseline, 3,6 and 12 months
  Headache Impact Test
Disability Measure | Baseline, 3,6 and 12 months
  Migraine Disability Assessment Score

OTHER OUTCOMES:
Abortive Medication Use | Through study completion
  Headache Diary

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's / Faulkner Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT06795867/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT06795867/ICF_001.pdf